CLINICAL TRIAL: NCT01951677
Title: Phase 1 Randomized, Controlled, Double-blind Study to Compare the Safety and Effectiveness of Hepatitis B Vaccines in Individuals With Renal Impairment, Diabetes Mellitus or Age Greater Than 40 Years
Brief Title: Safety and Efficacy Study of Adjuvanted Prophylactic Hepatitis B Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxine Pty Ltd (Industry)
Collaborators: Flinders Medical Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HBV002
Record Dates: First submitted 2013-09-16; First posted 2013-09-27 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Exposure to Hepatitis B Virus
Keywords: hepatitis B virus; vaccine; adjuvant; prophylaxis
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Surface Antigens; aluminum sulfate; Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- HBsAg + alum adjuvant (Active Comparator): HBsAg + standard alum adjuvant
  Interventions: Drug: HBsAg; Biological: Alum
- HBsAg + Advax-1(TM) (Experimental): HBsAg + Advax-1
  Interventions: Drug: HBsAg; Biological: Advax-1(TM)
- HBsAg + Advax-2(TM) (Experimental): HBsAg + Advax-2
  Interventions: Drug: HBsAg; Biological: Advax-2(TM)
- HBsAg + Advax-3(TM) (Experimental): HBsAg + Advax-3
  Interventions: Drug: HBsAg; Biological: Advax-3(TM)
- preS HBsAg + alum adjuvant (Active Comparator): preS HBsAg + alum adjuvant
  Interventions: Biological: PreS HBsAg; Biological: Alum
- preS HBsAg + Advax-1(TM) (Experimental): preS HBsAg + Advax-1
  Interventions: Biological: PreS HBsAg; Biological: Advax-1(TM)
- preS HBsAg + Advax-2(TM) (Experimental): preS HBsAg + Advax-2
  Interventions: Biological: PreS HBsAg; Biological: Advax-2(TM)
- preS HBsAg + Advax-3(TM) (Experimental): preS HBsAg + Advax-3
  Interventions: Biological: PreS HBsAg; Biological: Advax-3(TM)
- high dose preS HBsAg + alum adjuvant (Active Comparator): high dose preS HBsAg + alum adjuvant
  Interventions: Biological: PreS HBsAg; Biological: Alum
- high dose preS HBsAg + Advax-1(TM) (Experimental): high dose preS HBsAg + Advax-1
  Interventions: Biological: PreS HBsAg; Biological: Advax-1(TM)
- high dose preS HBsAg + Advax-2(TM) (Experimental): high dose preS HBsAg + Advax-2(TM)
  Interventions: Biological: PreS HBsAg; Biological: Advax-2(TM)
- high dose preS HBsAg + Advax-3(TM) (Experimental): high dose preS HBsAg + Advax-3
  Interventions: Biological: PreS HBsAg; Biological: Advax-3(TM)

INTERVENTIONS:
Drug: HBsAg — Standard hepatitis B vaccine antigen
  Other Names: hepatitis B vaccine based on hepatitis B surface antigen
  Arms: HBsAg + Advax-1(TM); HBsAg + Advax-2(TM); HBsAg + Advax-3(TM); HBsAg + alum adjuvant
Biological: PreS HBsAg — preS hepatitis B surface antigen
  Other Names: preS hepatitis B surface antigen
  Arms: high dose preS HBsAg + Advax-1(TM); high dose preS HBsAg + Advax-2(TM); high dose preS HBsAg + Advax-3(TM); high dose preS HBsAg + alum adjuvant; preS HBsAg + Advax-1(TM); preS HBsAg + Advax-2(TM); preS HBsAg + Advax-3(TM); preS HBsAg + alum adjuvant
Biological: Advax-1(TM) — Adjuvant formulated with vaccine antigen
  Other Names: Delta inulin adjuvant
  Arms: HBsAg + Advax-1(TM); high dose preS HBsAg + Advax-1(TM); preS HBsAg + Advax-1(TM)
Biological: Advax-2(TM) — Adjuvant formulated with vaccine antigen
  Other Names: Supermix
  Arms: HBsAg + Advax-2(TM); high dose preS HBsAg + Advax-2(TM); preS HBsAg + Advax-2(TM)
Biological: Advax-3(TM) — Adjuvant formulated with vaccine antigen
  Arms: HBsAg + Advax-3(TM); high dose preS HBsAg + Advax-3(TM); preS HBsAg + Advax-3(TM)
Biological: Alum — Adjuvant formulated with vaccine antigen
  Other Names: Alhydrogel; Aluminium hydroxide
  Arms: HBsAg + alum adjuvant; high dose preS HBsAg + alum adjuvant; preS HBsAg + alum adjuvant

SUMMARY:
There is a need for more effective and better-tolerated hepatitis B vaccines for low responder high-risk populations including patients with renal impairment and/or diabetes mellitus and those aged over 40 years. Several approaches are available to enhance the potency of hepatitis B virus vaccines including use of the more highly immunogenic antigens, replacing alum with potentially more effective adjuvants, and increasing the dose of vaccine antigen. A combination of these strategies is being tested in this study to identify the most promising candidate approaches to take forward into advanced clinical development

DETAILED DESCRIPTION:
Adjuvants are a critical ingredient in most vaccines and act by boosting the immune response to the target protein (e.g. hepatitis B surface antigen (HBsAg)). Despite considerable research, aluminium hydroxide or phosphate compounds (collectively referred to as "alum") remain the dominant adjuvants used in human hepatitis B virus vaccines. There is thus an unmet need for new HBV vaccine adjuvants, in particular, for adjuvants capable of boosting cell-mediated immunity (this is a particular type of immune response where killer T cells are activated that are then able to attack and destroy the infection) as alum, although good at stimulating antibodies is very poor at stimulating cell-mediated immunity. Alum, whilst generally accepted as safe, can be associated with significant local vaccine reactions and this is another reason why newer better-tolerated vaccine adjuvants would be beneficial. This study will compare a range of experimental adjuvant formulations to identify those that provide the safest and most effective enhancement of T- and B-cell immunity against hepatitis B

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Male or female
* Able to provide written informed consent
* Willing and able to comply with the protocol for the duration of the study.
* Has one or more of
* Age 40 years or above
* Impaired renal function (creatinine >120 mmol/L or calculated glomerular filtration rate <60mls/min)
* Diagnosis of diabetes mellitus (any type)

Exclusion Criteria:

* History of prior hepatitis B vaccination
* History of serious vaccine allergy if in the opinion of the Investigator this represents a contraindication to hepatitis B vaccination
* Women of childbearing potential unless using a reliable and appropriate contraceptive method, specifically oral contraceptive pill, intrauterine device or mechanical barrier device.
* Pregnant or lactating women.
* History of systemic autoimmune disease including Wegener's granulomatosis, systemic lupus erythematosus, Guillain-Barre, scleroderma or multiple sclerosis.
* Participation in another clinical trial with an investigational agent within 28 days of the scheduled date of first immunization.
* Any other serious medical, social or mental condition that, in the opinion of the investigator, would be detrimental to the subjects or the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Safety | 12 months
  Safety as assessed by incidence of adverse events

SECONDARY OUTCOMES:
Hepatitis B surface antibody geometric mean titer | one-month post each immunization and 10 months post-final immunization
  Geometric mean titer of HBsAg titers
T cell responses | 7 days and one month post each immunization and 10 months post-final immunization
  HBsAg-specific T cell responses as measured by cytokine enzyme-linked immunospot and carboxyfluorescein diacetate succinimidyl ester T-cell proliferation assay will be compared between groups
Efficacy | one month post each immunization and 10 months post final immunization
  Seroconversion and seroprotection rates will be compared between groups using titers of antibodies to hepatitis B surface antigen at each major time point

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Barbara, MBBS PhD, Principal Investigator — Flinders Medical Centre
Locations (1):
- Flinders Medical Centre, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
Currently no plan